CLINICAL TRIAL: NCT00248014
Title: Cephalometric Indicators of Biological Responsiveness to Orthodontic Treatment of Class II/I in Growing Patients
Brief Title: Response of Individuals With Class II Malocclusion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, IOANNA GIDARAKOU, Dr Ioanna Gidarakou, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORTHODONTICS 1
Record Dates: First submitted 2005-11-01; First posted 2005-11-03 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: CLASS II DIVISION 1 MALOCCLUSION
Keywords: CLASS II; FUNCTIONAL APPLIANCE; MANDIBULAR ADVANCEMENT STABILITY
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Mandibular Advancement Via A Functional Appliance — Functional appliance

SUMMARY:
This investigation aims at distinguishing the subjects that react in a favorable way to the treatment protocol we propose for the Class II treatment

DETAILED DESCRIPTION:
Class II Division 1 is a prevalent malocclusion. Many methods have been utilized to correct it.

The purpose of our prospective study is to clarify the specific cephalometric indicators of biological responsiveness that lead to a successful Class II Div.1 treatment in growing individuals. These indicators will hopefully assist in the differential diagnosis of a "true" and a "pseudo" Class II, that is a masked Class I, that we presume will be relatively easy to treat and stable a treatment result.

70 -100 subjects with a Class II/I malocclusion will be recruited and treated with the exact mode of treatment. As Class II we consider the one that is a t least half molar cusp Class II. Patients will already erupted lower first premolars will be included as we presume this is the approximate time of the maximum growth spurt which we want to exploit using the functional appliance. Crowding in both arches should not exceed 4 mm so as to exclude any denoalveolar changes due to alignment. Any tooth agenesis, besides the third molars, will exclude the subject from the study. The medical history of the patient should be non-contributory regarding any hormonal abnormalities, arthritis and pain from the TMJ. Syndromic patients and those exhibiting craniofacial abnormalities will be excluded.

The skeletal age of each patient will be assessed by observing the cervical column.

Every patient will have his records taken, the latter including a lateral ceph and a panoramic x-ray. Standard intra- and extra oral pictures will be taken as well (T0).

The treatment protocol includes a first phase of 3-4 months of slow palatal expansions utilizing a removable palatal plate with a 0.25 mm jackscrew in the middle (T1). The screw will be turned once a week for two weeks and then twice a week until the upper posterior teeth are over-expanded 2 mm per side. During phase II (T2)the patient will be asked to wear the same appliance adjusted as such to incorporate a tongue crib that will force the mandible into a Class I relationship acthing the way the know functional appliances work (eg activator). The crib will incorporate 4 loops in the canine area and will be placed so as not to impinge in the lower lingual gingival region but it will be long enough so as the patient will not be able to shift the mandible back. If the initial overjet exceeds 5 mm the mandibular advancement will be gradual. Further adjustments will be made so as to maintain the Class I relationship. The patient will wear the appliance for 8-12 months (T3). New records will be taken at that time. If braces are needed, the patient will continue with fixed appliances.

ELIGIBILITY:
Inclusion Criteria:

* Class II Division 1 malocclusion
* Crowding no more than 4 mm per side
* Healthy subjects

Exclusion criteria:

* Hormonal imbalances
* TMJ symptoms
* Craniofacial abnormalities
* Arthritis

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2005-10; Primary Completion 2008-11 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Achievement of Class I relationship | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: EFFI BASDRA, PHD, Study Director — ASSISTANT PROFESSOR
Locations (1):
- Orthodontic Clinic of Auth, Thessaloniki, Macedonia, Greece